CLINICAL TRIAL: NCT06091800
Title: Determination of Levels of IL-20, TNF-α, IL1β/IL-10, RANKL/OPG and MMP8 in Serum and Gingival Crevicular Fluid (GCF) in Peridontally Healthy and Periodontitis Individuals
Brief Title: Interleukin 20 and Periodontal Tisuue Destruction
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Hatice Yemenoglu, assistant professor, Recep Tayyip Erdogan University
Other Study IDs: RecepTayyip ErdoganUniversity; Recep Tayyip ErdoganUniversity (Other: Recep Tayyip Erdogan University)
Record Dates: First submitted 2023-10-11; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Biospecimen Retention: Samples With DNA — serum and gingival crevicular fluid
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group (periodontally healthy): no attachment loss, probing pocket depth ≤ 3 mm, minimal bleeding on probing ≤ 10%, and no radiographic bone loss
  Interventions: Other: biochemical analysis
- periodontitis group: interdental clinical attachment level ≥ 5 mm, probing pocket depth ≥ 6 mm, radiographic bone loss extending to the middle or apical thirds of the root, mid-crest defect, and a history of ≤4 teeth loss of periodontal origin
  Interventions: Other: biochemical analysis

INTERVENTIONS:
Other: biochemical analysis — GCF and serum samples were collected from the participants for biochemical analysis.

SUMMARY:
Periodontitis is an inflammatory disease that causes destruction of periodontal tissues. IL-20, on the other hand, is known as a potent angiogenic, chemotactic, and pro-inflammatory cytokine associated with various chronic inflammatory disorders. IL-20 has a significant role in the regulation of osteoclastogenesis and osteoblastogenesis. The aim of this study was to evaluate the effect of IL-20 on periodontal destruction.

In the study, a total of 60 participants were included, 30 of whom were systemically and periodontally healthy (control group) and 30 of whom were systemically healthy and had periodontitis (periodontitis group). GCF and serum samples were collected from the participants for biochemical analysis. ELISA method was used to determine IL-20, TNF-α, IL1β/IL-10, RANKL/OPG and MMP8 levels

ELIGIBILITY:
Inclusion Criteria:

* The following criteria were required for inclusion: being systemically healthy, not smoking, not using antibiotics or systemic corticosteroids within the previous three months, not being pregnant or nursing, not having a chronic inflammatory disease, not receiving periodontal therapy within the previous six months, and possessing at least 20 teeth

Exclusion Criteria:

* smoking, using antibiotics or systemic corticosteroids within the previous three months, pregnant, receiving periodontal therapy within the previous six months

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study included individuals who applied to Recep Tayyip Erdogan University, Faculty of Dentistry, Department of Periodontology for treatment
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
concentration of biochemical findings in gingival crevicular fluid (GCF) | june 2022-june 2023
  IL-20, RANKL, OPG and RANKL/OPG values eveluated in GCF
concentration of biochemical findings in serum | 1 year
  IL-20, RANKL, OPG, RANKL/OPG, MMP-8, TNF-α, IL-1β, IL-10 and IL-1β/IL-10

SECONDARY OUTCOMES:
value of periodontal clinical parameters | 1 year
  plaque index (PI) (Silness & Löe), gingival index (GI) (Silness & Löe) and bleeding on probing index (BOP) of all natural teeth of the patients
value of periodontal clinical parameters were measured in mm | 1 year
  probing pocket depth (PPD), clinical attachment loss (CAL) of all natural teeth of the patients

CONTACTS AND LOCATIONS:
Overall Officials: Yemenoglu, Principal Investigator — Recep Tayyip Erdogan University
Locations (1):
- Recep Tayyip Erdogan University, Rize, Turkey (Türkiye)